CLINICAL TRIAL: NCT00361569
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled Trial to Compare the Effects of 12 Weeks of Treatment With DR-2041(Synthetic Conjugated Estrogens, A) Vaginal Cream vs. Placebo Vaginal Cream on Vulvovaginal Atrophy in Healthy Postmenopausal Women
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of DR-2041(Synthetic Conjugated Estrogens, A) for Treatment of Vulvovaginal Atrophy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc.
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-CEN-302
Record Dates: First submitted 2006-08-03; First posted 2006-08-08 (Estimated); Results first posted 2009-04-14 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-03

CONDITIONS: Menopause
Keywords: vaginal atrophy; vaginal dryness; vaginal itching; vaginal pain
MeSH Terms: interventions — estrogens, conjugated synthetic A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: DR-2041a
- 2 (Experimental)
  Interventions: Drug: DR-2041b
- 3 (Placebo Comparator)
  Interventions: Other: Placebo
- 4 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DR-2041a — 1 gram administered vaginally daily for the 1st 7 days then twice a week thereafter
  Other Names: Synthetic conjugated estrogens, A
  Arms: 1
Drug: DR-2041b — 2 grams administered vaginally daily for the 1st 7 days then twice a week thereafter
  Other Names: Synthetic conjugated estrogens, A
  Arms: 2
Other: Placebo — 1 gram administered vaginally daily for the 1st 7 days then twice a week thereafter
  Arms: 3
Other: Placebo — 2 grams administered vaginally daily for the 1st 7 days then twice a week thereafter
  Arms: 4

SUMMARY:
This is a four-arm, randomized, double-blind, parallel group, placebo-controlled study to compare the effects of two doses of DR-2041(Synthetic Conjugated Estrogens, A) Vaginal Cream on vulvovaginal atrophy in postmenopausal women with or without a hysterectomy and/or oophorectomy.

DETAILED DESCRIPTION:
The study will include a screening period up to 4 weeks and a 12- week treatment period. The overall study duration for participants will be approximately 16 weeks. Study participants will undergo physical and gynecological exams, and blood tests for clinical laboratory assessments. All patients with a uterus will undergo transvaginal ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Naturally or surgically menopausal
* Moderate or severe symptoms of vaginal atrophy (ie, dryness, itching, pain, uncomfortable intercourse)

Exclusion Criteria:

* Known sensitivity or contraindication to estrogens or progestins
* History or current diagnosis endometrial hyperplasia
* Recent history of vaginal bleeding of unknown cause
* Recent history or diagnosis of endometriosis
* Any contraindication to estrogen therapy

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (80):
- United States (80):
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Mobile, Alabama
  - Duramed Investigational Site, Montgomery, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Carmichael, California
  - Duramed Investigational Site, Fresno, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, San Ramon, California
  - Duramed Investigational Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Pueblo, Colorado
  - Duramed Investigational Site, New London, Connecticut
  - Duramed Investigational Site, Clearwater, Florida
  - Duramed Investigational Site, Gainesville, Florida
  - Duramed Investigational Site, Jacksonville, Florida
  - Duramed Investigational Site, Leesburg, Florida
  - Duramed Investigational Site, Miami, Florida
  - Duramed Investigational Site, Pinellas Park, Florida
  - Duramed Investigational Site, Stuart, Florida
  - Duramed Investigational Site, Tampa, Florida
  - Duramed Investigational Site, Venice, Florida
  - Duramed Investigational Site, West Palm Beach, Florida
  - Duramed Investigational Site, Weston, Florida
  - Duramed Investigational Site, Alpharetta, Georgia
  - Duramed Investigational Site, Atlanta, Georgia
  - Duramed Investigational Site, Augusta, Georgia
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Investigational Site, Douglasville, Georgia
  - Duramed Investigational Site, Sandy Springs, Georgia
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Evansville, Indiana
  - Duramed Investigational Site, Overland Park, Kansas
  - Duramed Investigational Site, Lexington, Kentucky
  - Duramed Investigational Site, Louisville, Kentucky
  - Duramed Investigational Site, Madisonville, Kentucky
  - Duramed Investigational Site, Shreveport, Louisiana
  - Duramed Investigational Site, Baltimore, Maryland
  - Duramed Investigational Site, Livonia, Michigan
  - Duramed Investigational Site, Lincoln, Nebraska
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Lebanon, New Hampshire
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, New Brunswick, New Jersey
  - Duramed Investigational Site, Albuquerque, New Mexico
  - Duramed Investigational Site, Johnson City, New York
  - Duramed Investigational Site, Williamsville, New York
  - Duramed Investigational Site, Raleigh, North Carolina
  - Duramed Investigational Site, Winston-Salem, North Carolina
  - Duramed Investigational Site, Jamestown, North Dakota
  - Duramed Investigational Site, Minot, North Dakota
  - Duramed Investigational Site, Cincinnati, Ohio
  - Duramed Investigational Site, Cleveland, Ohio
  - Duramed Investigational Site, Columbus, Ohio
  - Duramed Investigational Site, Mayfield Heights, Ohio
  - Duramed Investigational Site, Medford, Oregon
  - Duramed Investigational Site, Portland, Oregon
  - Duramed Investigational Site, Allentown, Pennsylvania
  - Duramed Investigational Site, King of Prussia, Pennsylvania
  - Duramed Investigational Site, Media, Pennsylvania
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Rosemont, Pennsylvania
  - Duramed Investigational Site, Strafford, Pennsylvania
  - Duramed Investigational Site, Warwick, Rhode Island
  - Duramed Investigational Site, Charleston, South Carolina
  - Duramed Investigational Site, Columbia, South Carolina
  - Duramed Investigational Site, Watertown, South Dakota
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Nashville, Tennessee
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Corpus Christi, Texas
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Waco, Texas
  - Duramed Investigational Site, Williston, Vermont
  - Duramed Investigational Site, Newport News, Virginia
  - Duramed Investigational Site, Spokane, Washington
  - Duramed Investigational Site, Tacoma, Washington

REFERENCES:
- [Result] Freedman M, Kaunitz AM, Reape KZ, Hait H, Shu H. Twice-weekly synthetic conjugated estrogens vaginal cream for the treatment of vaginal atrophy. Menopause. 2009 Jul-Aug;16(4):735-41. doi: 10.1097/gme.0b013e318199e734. PMID 19252451

RESULTS

PARTICIPANT FLOW:
Groups:
- DR-2041a: Synthetic Conjugated Estrogens, A (DR-2041)-1 gram administered vaginally daily for the 1st 7 days then twice a week thereafter
- DR-2041b: Synthetic Conjugated Estrogens, A (DR-2041)-2 grams administered vaginally daily for the 1st 7 days then twice a week thereafter
- Placebo-a: 1 gram administered vaginally daily for the 1st 7 days then twice a week thereafter
- Placebo-b: 2 grams administered vaginally daily for the 1st 7 days then twice a week thereafter
Period: Overall Study
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Started | 150 | 161 | 155 | 156
Completed | 138 | 150 | 137 | 135
Not Completed | 12 | 11 | 18 | 21
Not completed — Protocol Violation | 3 | 2 | 4 | 2
Not completed — Withdrawal by Subject | 2 | 1 | 9 | 14
Not completed — Adverse Event | 3 | 5 | 2 | 2
Not completed — Lost to Follow-up | 2 | 3 | 3 | 2
Not completed — Not specified by investigator | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b | Total
Number analyzed (Participants) | 150 | 161 | 155 | 156 | 622
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (6.48) | 59.3 (6.10) | 59.8 (6.60) | 58.4 (6.28) | 59.4 (6.36)
Age, Customized [Number; unit: participants]
  Between 30 and 80 years | 150 | 161 | 155 | 156 | 622.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150 | 161 | 155 | 156 | 622.0
  Male | 0 | 0 | 0 | 0 | 0.0
Region of Enrollment [Number; unit: participants]
  United States | 150 | 161 | 155 | 156 | 622.0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in the Symptom Identified by the Patient to be Most Bothersome
Description: Change= Week 12 score - Baseline Score. The most bothersome symptom was derived from the subject self-assessment of vaginal atrophy, which consisted of 5 questions concerning severity of symptoms graded on a scale of 0-3(none, mild, moderate or severe) or 7 for not applicable.
Time Frame: Baseline to Week 12
Population: Modifed Intent-to-Treat: All subjects meeting study protocol requirements at baseline for all 3 primary efficacy inclusion criteria, randomized to treatment, received at least 1 dose of study drug, and had a baseline assessment and at least 1 post-randomization assessment of vulvovaginal atrophy consisting of all 3 co-primary efficacy endpoints
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Number analyzed (Participants) | 135 | 146 | 140 | 135
Scores on a scale | -1.71 (0.0087) | -1.77 (0.085) | -1.11 (0.086) | -1.10 (0.087)

2. Primary Outcome: Mean Change in Vaginal pH
Description: Change= Week 12 vaginal pH - Baseline vaginal pH
Time Frame: Baseline to Week 12
Population: Modifed Intent-to-Treat: All subjects who met study protocol requirements at baseline for all 3 primary efficacy inclusion criteria, who were randomized to treatment, received at least 1 dose of study drug, for whom there were a baseline assessment and at least 1 post-randomization assessment of VVA consisting of all 3 co-primary efficacy endpoints
Measure: Least Squares Mean (Standard Error); unit: pH
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Number analyzed (Participants) | 135 | 146 | 140 | 135
pH | -1.48 (0.073) | -1.44 (0.071) | -0.31 (0.072) | -0.38 (0.073)

3. Primary Outcome: Mean Change in Maturation Index
Description: Change= Week 12 maturation index -baseline maturation index. Matuation index was calculated using the following equation: Maturation Index = (% Parabasal cells * 0) + (% Intermediate Cells * 0.5) + (% Superficial Cells * 1.0)
Time Frame: Baseline to Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Index
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Number analyzed (Participants) | 135 | 146 | 140 | 135
Index | 31.46 (1.221) | 33.27 (1.191) | 5.16 (1.205) | 8.91 (1.222)

4. Secondary Outcome: Safety and Tolerability of DR-2041 (Synthetic Conjugated Estrogens, A)
Description: Any adverse event reported from the beginning of the 28-day screening through the subject's last report.
Time Frame: Up to Week 12
Population: All randomized subjects who received at least one dose of study medication
Measure: Number; unit: Participants
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Number analyzed (Participants) | 150 | 161 | 155 | 156
Participants | 83 | 87 | 72 | 77

ADVERSE EVENTS:
Time Frame: Adverse event reporting began on the first day of signing the informed consent and ended at the end of study drug treatment (approximately 16 weeks).
Description: Adverse events were reported during the subject's regularly scheduled visits at the investigational site. Adverse events reported are those that emerged during the treatment period.
Arm/Group | DR-2041a | DR-2041b | Placebo-a | Placebo-b
Serious Adverse Events (participants affected / at risk) | 1/150 | 1/161 | 1/155 | 3/156
Other Adverse Events (participants affected / at risk) | 34/150 | 36/161 | 18/155 | 33/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-2041a (N=150) | DR-2041b (N=161) | Placebo-a (N=155) | Placebo-b (N=156)
Cardiac Chest Pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic Sinusitus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DR-2041a (N=150) | DR-2041b (N=161) | Placebo-a (N=155) | Placebo-b (N=156)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 7 (7) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 0 (0) | 2 (2)
Genital Pruritus Female (Reproductive system and breast disorders) | 4 (4) | 5 (5) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 6 (6)
Hot Flush (Vascular disorders) | 5 (5) | 2 (2) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7) | 6 (6) | 7 (7) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 5 (5) | 2 (2) | 6 (6)
Vulvovaginal Mycotic Infection (Infections and infestations) | 7 (7) | 3 (3) | 5 (5) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can (i) review results communications prior to public release and can embargo communications regarding trial results for a period of at least 60 days but no more than 180 days from the time submitted to the sponsor for review; and (ii) require in instances of a multi-center study, that a single PI not disclose study data until after the multi-center results are published, provided such results are published within eighteen (18) months of the conclusion of the study.